CLINICAL TRIAL: NCT05673603
Title: A Phase 1, Open-Label, Single Dose Parallel-Group Study of Brensocatib Following a Single Oral Administration in Subjects With or Without Renal Impairment
Brief Title: A Study of Brensocatib Following a Single Oral Administration in Participants With or Without Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS1007-102
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Renal Impairment
Keywords: Brensocatib; INS1007
MeSH Terms: conditions — Renal Insufficiency | interventions — brensocatib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Mild Impairment): Brensocatib (Experimental): Participants with mild renal impairment will receive single oral dose of brensocatib on Day 1 under fasted conditions.
  Interventions: Drug: Brensocatib
- Cohort 2 (Moderate Impairment): Brensocatib (Experimental): Participants with moderate renal impairment will receive single oral dose of brensocatib on Day 1 under fasted conditions.
  Interventions: Drug: Brensocatib
- Cohort 3 (Severe Impairment): Brensocatib (Experimental): Participants with severe renal impairment will receive single oral dose of brensocatib on Day 1 under fasted conditions.
  Interventions: Drug: Brensocatib
- Cohort 4 (Normal): Brensocatib (Experimental): Healthy participants with normal renal function will receive single oral dose of brensocatib on Day 1 under fasted conditions. Healthy participants will be matched within the protocol criteria to one or more participants with renal impairment.
  Interventions: Drug: Brensocatib

INTERVENTIONS:
Drug: Brensocatib — Oral tablet
  Other Names: INS1007

SUMMARY:
The primary purpose of the study is to determine the pharmacokinetics (PK) following a single oral dose administration of brensocatib, safety, and tolerability of brensocatib when administered to participants with impaired renal function and in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) 18 to 35 kilograms per square meter (kg/m^2), inclusive, and a body weight of ≥50 kg at Screening.

Inclusion Criteria (for Participants With Renal Impairment):

* Mild, moderate, or severe renal impairment as determined by estimated glomerular filtration rate (eGFR) and calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
* Renal insufficiency or other related concomitant medical conditions (e.g., hypertension, anemia) has remained stable for at least 3 months before study drug dosing.

Inclusion Criteria for Healthy Participants:

* Normal renal function as determined by eGFR and calculated using the CKD-EDI formula, or by 24-hour urine creatinine clearance (CLcr) corrected for body size.
* In good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12-lead electrocardiogram (ECG) results, and physical examination findings.

Exclusion Criteria:

* Positive test result for human immunodeficiency virus types 1 or 2 antibodies, hepatitis C virus antibodies, or hepatitis B surface antigen or hepatitis B core antibodies.
* History of relevant drug and/or food allergies (i.e., allergy to brensocatib or any excipients, or any significant food allergy).
* The participant has received study drug in another investigational study within 30 days of Screening.

Exclusion Criteria (for Participants With Renal Impairment):

* Has nephrotic syndrome, defined as urine dipstick 4+ for protein and plasma albumin <3.0 grams per deciliter (g/dL), and then confirmed if proteinuria >5 g/day.
* Has an extrarenal cause of renal impairment (e.g., rapidly growing, space occupying lesions, adrenal enlargement).
* Has a functioning renal transplant (participant may be included in the study if he or she had a failed renal transplant and is not taking immunosuppressants).
* Has a hemoglobin value less than 8.5 g/dL.
* Has Type 1 or Type 2 diabetes mellitus.

Exclusion Criteria (for Healthy Participants):

* Has used any prescription (excluding hormonal birth control, hormone replacement therapy, nonsteroidal anti-inflammatory drugs, or acetaminophen) or over-the-counter medications, including herbal or nutritional supplements, within 14 days before study drug dosing and throughout the study.

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Time Curve (AUC) of Brensocatib | Pre-dose and at multiple timepoints post-dose on Days 1 to 14
  Pharmacokinetics of brensocatib following a single dose will be assessed in participants with renal impairment and in healthy participants.
Maximum Observed Plasma Concentration (Cmax) of Brensocatib | Pre-dose and at multiple timepoints post-dose on Days 1 to 14
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Brensocatib | Pre-dose and at multiple timepoints post-dose on Days 1 to 14
Number of Participants who Experienced at Least one Adverse Event (AE) | Up to Day 14
  Determination of the safety and tolerability of a single dose of brensocatib in participants with impaired renal function and in healthy participants.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - USA002, Orlando, Florida
  - USA003, Tampa, Florida
  - USA001, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeung SA, Stein DS, Marbury TC, Usansky H. The pharmacokinetics of brensocatib in participants with renal impairment following a single oral administration. Br J Clin Pharmacol. 2025 Apr;91(4):1191-1197. doi: 10.1111/bcp.16344. Epub 2024 Nov 22. PMID 39574348